CLINICAL TRIAL: NCT06198439
Title: Higher Neural and Clinical Effects of Non-Invasive Transcranial Neuromodulation in Adults With Overactive Bladder
Brief Title: rTMS in Overactive Bladder
Acronym: TMS_OAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRO00037607
Record Dates: First submitted 2023-10-02; First posted 2024-01-10 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Overactive Bladder; Overactive Bladder Syndrome; Urge Incontinence; Urgency-frequency Syndrome; Urinary Incontinence; Urinary Incontinence, Urge
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urinary Incontinence | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Prospective cohort study, all subjects receive the same intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Transcranial magnetic stimulation (Experimental): All study subjects undergo five sessions of rTMS. The 40-minute sessions target the supplemental motor area (inhibitory stimulation) and prefrontal cortex (excitatory stimulation)
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Magstim Rapid2 Therapy System
  Other Names: Magstim Rapid2 Therapy System

SUMMARY:
Overactive bladder (OAB) imposes a significant quality of life, mental health, and economic burdens. OAB with or without Urgency incontinence is associated with depression, sexual dysfunction, and limitation of social interactions and physical activities, which significantly affects quality of life.

Non-invasive neuromodulation with repetitive transcranial magnetic stimulation (rTMS) can be used in research settings to investigate responses to focal regional brain activation. In the clinical setting, rTMS normalizes brain activity with associated clinical benefits in conditions such as refractory depression. rTMS has been studied for effects on lower urinary tract symptoms (LUTS) in bladder pain and neurogenic lower urinary tract symptoms (LUTS) populations.

Unlike many standard of care OAB interventions, the safety of rTMS is well-reported, including for use in elderly populations and those with cognitive impairment. Functional magnetic resonance imaging (fMRI) to evaluate neuroplasticity is emerging as an essential tool to define OAB phenotypes; however, phenotyping studies guided by mechanistic data are lacking. The effects of central neuromodulation on regions involved OAB mechanisms and associated physiological and clinical responses are unknown. This study will be the first to report neuroplasticity, physiologic, and clinical effects of central neuromodulation with rTMS in adults with OAB.

DETAILED DESCRIPTION:
This prospective trial will enroll eligible adults with OAB recruited from Urology and urogynecology clinics. Subjects have a baseline evaluation with questionnaires, clinical data, and fMRI to assess brain activity during urinary urgency. All subjects receive the intervention: 5 daily sessions of rTMS to regions of interest. Electromyography will assess pelvic floor muscle activity at rest during rTMS. Following the intervention, an evaluation with questionnaires, clinical data, and fMRI is repeated.

ELIGIBILITY:
Inclusion Criteria:

* Females & Males
* 40 to 80 years old
* 3 months of OAB symptoms without active urinary tract infection currently
* Bladder diary:

  * Mean voids/24 hours ≥ 8.0
  * Mean urgency episodes/24 hours ≥ 3.0
* Montreal Cognitive Assessment (MoCA) score >10

Exclusion Criteria:

* Pregnant, nursing, or self-report of planning to become pregnant.
* Contraindication to MRI or to the Rapid2 Magstim Device as listed in the operator manual
* Qmax < 10 ml/s in males on uroflow
* < 20th percentile on Liverpool nomogram
* Postvoid residual volume ≥ 200 mL, suprapubic or indwelling catheter
* Personal or immediate family history of seizure disorder
* Taking (bupropion) Wellbutrin or heavy alcohol use
* Parkinson's disease, Multiple sclerosis, spinal cord injury
* Intracranial lesions and hemorrhagic stroke within the last 12 months
* History of interstitial cystitis, pelvic radiation, bladder augmentation
* Intradetrusor botulinum toxin injections within 6 months
* Pelvic floor therapy within 2 months.
* Active/on-mode Sacral nerve stimulator (eligible if turned off)
* Incarcerated patients

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Regional brain activity | Post-intervention at: 0 to 3 days
  Activity in the supplemental motor area and prefrontal cortex during full bladder
Functional connectivity | Post-intervention at: 0 to 3 days
  Connectivity of regions of interest with a full bladder and empty bladder state

SECONDARY OUTCOMES:
Pelvic floor muscle activity | on day 5 of the intervention
  Surface electromyography of the pelvic floor muscles during rTMS sessions with subjects at rest
Urinary frequency | Post-intervention at: 1 day, 3 weeks, 6 weeks
  Mean Voids per 24 hours (n) 2- day bladder diary (higher score is worse outcome)
Urgency episodes | Post-intervention at: 1 day, 3 weeks, 6 weeks
  Mean urgency episodes per 24 hours (n) 2- day bladder diary (higher score is worse outcome)
OAB Symptom Bother | Post-intervention at: 1 day, 3 weeks, 6 weeks
  OAB-q symptom burden score (higher score is worse outcome)
OAB related Quality of life | Post-intervention at: 1 day, 3 weeks, 6 weeks
  OAB-q health-related quality of life score (higher score is a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Almarez, BBA, Study Director — Houston Methodist Obstetrics & Gynecology Department
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No